CLINICAL TRIAL: NCT02529995
Title: Phase I, Open-Label, Two Parts Study in Chinese Patients With Advanced NSCLC Who Have Progressed Following Prior Therapy With an EGFR Tyrosine Kinase Inhibitor Agent
Brief Title: Phase I, Study in Chinese NSCLC Patients
Acronym: AURAChinaPK
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: D5160C00018
Record Dates: First submitted 2015-08-06; First posted 2015-08-20 (Estimated); Results first posted 2017-03-06 (Actual); Last update posted 2020-02-11 (Actual); Status verified 2020-02

CONDITIONS: Carcinoma, Non-Small-Cell Lung With EGFR Mutation Positive
MeSH Terms: conditions — Carcinoma | interventions — osimertinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- AZD9291 40 mg (Experimental): Cohort 1: 40 mg once daily
  Interventions: Drug: AZD9291 40 mg
- AZD9291 80 mg (Experimental): Cohort 2: 80 mg once daily
  Interventions: Drug: AZD9291 80 mg

INTERVENTIONS:
Drug: AZD9291 40 mg — This is a two parts (Part A and Part B) study to determine the pharmacokinetics of AZD9291 administered orally at two dose levels (40 mg Cohort 1 and 80 mg Cohort 2) in patients with locally advanced or metastatic NSCLC who have progressed following prior therapy with an EGFR TKI agent (+/- additional chemotherapy regimens).
  Arms: AZD9291 40 mg
Drug: AZD9291 80 mg — This is a two parts (Part A and Part B) study to determine the pharmacokinetics of AZD9291 administered orally at two dose levels (40 mg Cohort 1 and 80 mg Cohort 2) in patients with locally advanced or metastatic NSCLC who have progressed following prior therapy with an EGFR TKI agent (+/- additional chemotherapy regimens).
  Arms: AZD9291 80 mg

SUMMARY:
A Phase I, Open-Label, Two Parts Study to Assess the Safety, Tolerability,Pharmacokinetics and Preliminary Anti-tumour Activity of AZD9291 in Chinese Patients with Advanced Non-Small Cell Lung Cancer who have Progressed Following Prior Therapy with an Epidermal Growth Factor Receptor Tyrosine Kinase Inhibitor Agent

Study Objective: 1, Primary Objective To characterise the pharmacokinetics (PK) of AZD9291 and its metabolites (AZ5104 and AZ7550) after single then multiple doses of AZD9291 administered orally once daily in Chinese patients with locally advanced or metastatic non small cell lung Cancer (NSCLC) who have progressed following prior therapy with an approved Epidermal Growth Factor Receptor Tyrosine Kinase Inhibitor (EGFR TKI) agent.

2, Secondary objective(s) To investigate the safety and tolerability of AZD9291 when given orally to Chinese patients with locally advanced or metastatic NSCLC who have progressed following prior therapy with an approved EGFR TKI agent. To obtain a preliminary assessment of the anti-tumour activity of AZD9291 by evaluation of tumour response using Response Evaluation Criteria in Solid Tumours (RECIST) version 1.1.

DETAILED DESCRIPTION:
This is a phase I, open-label, two parts (Part A and Part B) study to determine the pharmacokinetics of AZD9291 administered orally at two dose levels (40 mg and 80 mg) in patients with locally advanced or metastatic NSCLC who have progressed following prior therapy with an approved EGFR TKI agent (+/- additional chemotherapy regimens).

Approximately 24 patients will enter into this study, with 12 patients at each dose level.

* Cohort 1 will investigate the pharmacokinetics of single then multiple dosing of AZD9291 at 40 mg once daily dose.
* Cohort 2 will investigate the pharmacokinetics of single then multiple dosing of AZD9291 at 80 mg once daily dose.

The enrollment of Cohort 2 will start after Cohort 1 finishes the enrollment. The first 12 patients enrolled in the study will be in 40 mg dose Cohort.

Patients will be administered a single dose of AZD9291 on Day 1, Cycle 0 at the beginning of Part A period. From Day 2 to Day 6, no treatment will be given, but PK samples will be obtained; on Day 7 (Cycle1, Day1), the patients will be administered AZD9291 once daily on a continuous schedule, ie, no break in AZD9291 dosing. Part A will complete after Cycle 4 treatment and Part B will start without treatment interruption.

Patients in both cohorts should continue on treatment with AZD9291 until a treatment discontinuation criterion is met. There is no maximum duration of treatment as patients may continue to receive AZD9291 beyond RECIST 1.1 defined progression as long as they are continuing to receive clinical benefit, as judged by the investigator.

The whole study will be divided nominally into two parts: Part A will assess the pharmacokinetics and preliminary efficacy and safety of AZD9291 at 40 mg and 80 mg respectively, and Part B will assess only the safety and efficacy data of AZD9291.

Following completion of the Part A, patients will automatically continue to Part B.

ELIGIBILITY:
Inclusion Criteria:

1. Provision informed consent
2. Aged at least 18 years
3. Histological or cytological confirmation diagnosis of NSCLC
4. Locally advanced or metastatic NSCLC
5. Radiological documentation of disease progression while on a previous continuous treatment with an approved EGFR TKI. In addition other lines of therapy may have been given

   * Documented EGFR mutation (at any time since the initial diagnosis of NSCLC) known to be associated with EGFR TKI sensitivity (including G719X, exon 19 deletion, L858R, L861Q)
6. World Health Organisation (WHO) performance status 0-1
7. At least one lesion suitable for accurate repeated measurements
8. Females

   * Child bearing potential : should not be breast feeding, use adequate contraceptive measures for female patients with child-bearing potential, OR
   * Have evidence of non-child-bearing potential that meet one of the following criteria at screening:
   * Post-menopausal defined as aged more than 50 years and amenorrhoeic for at least 12 months following cessation of all exogenous hormonal treatments
   * Women below 50 years old would be consider postmenopausal if they have been amenorrheic for 12 months or more following cessation of exogenous hormonal treatments and with luteinizing hormone (LH) and follicle-stimulating hormone (FSH) levels in the post-menopausal range for the institution
   * Documentation of irreversible surgical sterilisation by hysterectomy, bilateral oophorectomy or bilateral salpingectomy but not tubal ligation
9. Male patients should be willing to use barrier contraception ie, condoms

Exclusion Criteria:

1. Treatment with any of the following (prior to first dose of study treatment)

   * Treatment with an EGFR TKI within 8 days
   * Any investigational agents or other anticancer drugs from a previous treatment regimen or clinical study within 14 days
   * Previous treatment with AZD9291, or a Thr790Met (T790M) directed EGFR TKIs
   * Major surgery (excluding placement of vascular access) within 4 weeks
   * Radiotherapy :
   * Within 1 week if limited field of radiation for palliation of the first dose of study treatment
   * Within 4 weeks if receiving radiation to more than 30% of the bone marrow or with a wide field of radiation
   * Patients currently receiving (or unable to stop use at least 1 week) medications or herbal supplements known to be potent inhibitors or inducers of cytochrome P450 3A4 (CYP3A4)
   * Treatment with an investigational drug within five half-lives of the compound
2. Any unresolved toxicities from prior therapy greater than CTCAE grade 1 at the time of starting study treatment with the exception of alopecia and grade 2, prior platinum-therapy related neuropathy
3. Spinal cord compression or brain metastases unless asymptomatic, stable and not requiring steroids for at least 4 weeks prior to start of study treatment
4. Any evidence of severe or uncontrolled systemic diseases, including uncontrolled hypertension and active bleeding diatheses, which in the investigator's opinion makes it undesirable for the patient to participate in the trial or which would jeopardise compliance with the protocol, or active infection including hepatitis B, hepatitis C and human immunodeficiency virus (HIV). Screening for chronic conditions is not required
5. Any of the following cardiac criteria:

   * Mean resting corrected QT interval (QTc) >470 msec obtained from 3 electrocardiograms (ECGs), using the screening clinic ECG machine derivedQTc value
   * Any clinically important abnormalities in rhythm, conduction or morphology of resting ECG eg, complete left bundle branch block, third degree heart block, second degree heart block, P wave to R wave (PR) interval >250 msec
   * Any factors that increase the risk of QTc prolongation or risk of arrhythmic events such as heart failure, hypokalaemia, congenital long (Q-T interval) QT syndrome, family history of long QT syndrome or unexplained sudden death under 40 years of age in first degree relatives or any concomitant medication known to prolong the QT interval
6. Past medical history of interstitial lung disease, drug-induced interstitial lung disease, radiation pneumonitis which required steroid treatment, or any evidence of clinically active interstitial lung disease 7, Inadequate bone marrow reserve or organs function as demonstrated by any of the following laboratory values:

   * Absolute neutrophil count <1.5x109/L
   * Platelet count <100x109/L
   * Hemoglobin <90 g/L
   * Alanine aminotransferase >2.5 times the upper limit of normal (ULN) if no demonstrable liver metastases or >5 times ULN in the presence of liver metastases
   * Aspartate aminotransferase >2.5 times ULN if no demonstrable liver metastases or >5 times ULN in the presence of liver metastases
   * Total bilirubin >1.5 times ULN if no liver metastases or >3 times ULN in the presence of documented Gilbert's Syndrome (unconjugated hyperbilirubinaemia) or liver metastases
   * Creatinine >1.5 times ULN concurrent with creatinine

8, Clearance <50 ml/min (measured or calculated by Cockcroft and Gault equation); confirmation of creatinine clearance is only required when creatinine is >1.5 times ULN Refractory nausea and vomiting, chronic gastrointestinal diseases, inability to swallow the formulated product or previous significant bowel resection that would preclude adequate absorption of AZD9291 9, History of hypersensitivity to active or inactive excipients of AZD9291 or drugs with a similar chemical structure or class to AZD9291 10, Women who are breast feeding 11, Involvement in the planning and conduct of the study (applies to AstraZeneca staff or staff at the study site) 12, Judgement by the investigator that the patient should not participate in the study if the patient is unlikely to comply with study procedures, restrictions and requirements

Ages: 18 Years to 130 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2015-08-24 (Actual); Primary Completion 2016-01-28 (Actual); Study Completion 2019-09-27 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Research Site, Guangzhou
  - Research Site, Shanghai

REFERENCES:
- [Derived] Zhao H, Cao J, Chang J, Zhang Z, Yang L, Wang J, Cantarini M, Zhang L. Pharmacokinetics of Osimertinib in Chinese Patients With Advanced NSCLC: A Phase 1 Study. J Clin Pharmacol. 2018 Apr;58(4):504-513. doi: 10.1002/jcph.1042. Epub 2017 Dec 14. PMID 29239002
- See also: AURA18_Redacted — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=3753&filename=AURA18_Redacted.pdf

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All patients were enrolled in China: first patient enrolled on 24-08-2015. The recruitment was closed following LSI. The primary analysis for the PK was performed at the data cut off (DCO1): 28-01-2016. The study was on-going until the final analysis for the efficacy & safety at the data cut off (DCO2): 02-11-2016 and the study is completed.
Pre-assignment Details: 36 patients were enrolled (signed informed consent). Patients were assigned to treatment if they met all the inclusion and none of the exclusion criteria. 4 patients were enrolled but failed inclusion/exclusion criteria and 1 patient withdrew consent so were not eligible to be assigned treatment. The remaining 31 patients received treatment.
Groups:
- AZD9291 40mg: Single oral dose of AZD9291 40mg on Cycle 0 Day 1
- AZD9291 80mg: Single oral dose of AZD9291 80mg on Cycle 0 Day 1
Period: Part A
Arm/Group | AZD9291 40mg | AZD9291 80mg
Started | 15 | 16
Completed | 0 ('Completed' means 'Completed the Study', i.e. zero patient completed the study in part A.) | 0 ('Completed' means 'Completed the Study', i.e. zero patient completed the study in part A.)
Not Completed | 15 | 16
Not completed — Ongoing Study at Data Cut-off | 14 | 16
Not completed — Discontinued Study | 1 | 0
Period: Part B
Arm/Group | AZD9291 40mg | AZD9291 80mg
Started | 15 | 16
Completed | 9 | 4
Not Completed | 6 | 12
Not completed — Ongoing Study at Data Cut-off | 0 | 7
Not completed — Discontinued Study | 6 | 5

BASELINE CHARACTERISTICS:
Population: All patients enrolled who received at least one dose of AZD9291.
Groups:
- Total: Total of all reporting groups
Arm/Group | AZD9291 40mg | AZD9291 80mg | Total
Number analyzed (Participants) | 15 | 16 | 31
Age, Continuous [Mean (Standard Deviation); unit: Years] | 54.1 (10.78) | 60.1 (10.92) | 57.2 (11.10)
Age, Customized [Number; unit: Participants]
  <50 Years | 4 | 2 | 6
  >=50-<65 Years | 8 | 7 | 15
  >=65-<75 Years | 3 | 6 | 9
  >=75 Years | 0 | 1 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 11 | 18
  Male | 8 | 5 | 13
Race/Ethnicity, Customized [Number; unit: Participants]
  Asian/Chinese | 15 | 16 | 31

OUTCOME MEASURES:

1. Primary Outcome: Cmax of AZD9291 After Single Dosing
Description: Pharmacokinetics of AZD9291 after single dosing by assessment of maximum plasma AZD9291 concentration
Time Frame: PK blood samples are collected at pre-dose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 48, 72 and 120 hours post-dose. Results are based on data cut off of 28 Jan 2016.
Population: Pharmacokinetic population - all patients who received at least 1 dose of AZD9291 and had at least 1 quantifiable plasma concentration collected post-dose without important protocol deviations/violations. Overall number of participants analyzed is the number of patients in Pharmacokinetic population who had available data for each PK variable.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nmol/L
Arm/Group | AZD9291 40mg | AZD9291 80mg
Number analyzed (Participants) | 12 | 13
nmol/L | 103.8 (79.21) | 195.9 (49.83)

2. Primary Outcome: Cmax of AZ5104 After Single Dosing
Description: Pharmacokinetics of AZD9291 metabolites (AZ5104) after single dosing by assessment of maximum plasma concentration
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nmol/L
Arm/Group | AZD9291 40mg | AZD9291 80mg
Number analyzed (Participants) | 12 | 13
nmol/L | 4.207 (79.85) | 9.582 (71.63)

3. Primary Outcome: Cmax of AZ7550 After Single Dosing
Description: Pharmacokinetics of AZD9291 metabolites (AZ7550) after single dosing by assessment of maximum plasma concentration
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nmol/L
Arm/Group | AZD9291 40mg | AZD9291 80mg
Number analyzed (Participants) | 12 | 13
nmol/L | 3.443 (68.42) | 7.842 (50.62)

4. Primary Outcome: AUC of AZD9291 After Single Dosing
Description: Pharmacokinetics of AZD9291 after single dosing by assessment of area under the plasma concentration time curve from zero to infinity
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nmol*h/L
Arm/Group | AZD9291 40mg | AZD9291 80mg
Number analyzed (Participants) | 11 | 13
nmol*h/L | 6323 (55.81) | 10260 (33.10)

5. Primary Outcome: AUC of AZ5104 After Single Dosing
Description: Pharmacokinetics of AZD9291 metabolites (AZ5104) after single dosing by assessment of area under the plasma concentration time curve from zero to infinity
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nmol*h/L
Arm/Group | AZD9291 40mg | AZD9291 80mg
Number analyzed (Participants) | 7 | 12
nmol*h/L | 589.0 (74.20) | 1077 (57.22)

6. Primary Outcome: AUC of AZ7550 After Single Dosing
Description: Pharmacokinetics of AZD9291 metabolites (AZ7550) after single dosing by assessment of area under the plasma concentration time curve from zero to infinity
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nmol*h/L
Arm/Group | AZD9291 40mg | AZD9291 80mg
Number analyzed (Participants) | 5 | 5
nmol*h/L | 527.4 (46.61) | 1292 (29.31)

7. Primary Outcome: CL/F of AZD9291 After Single Dosing
Description: Rate and extent of absorption of single dose AZD9291 by assessment of apparent clearance following oral administration
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: L/h
Arm/Group | AZD9291 40mg | AZD9291 80mg
Number analyzed (Participants) | 11 | 13
L/h | 14.30 (7.701) | 16.45 (6.086)

8. Primary Outcome: C(ss, Max) of AZD9291 After Multiple Dosing
Description: Pharmacokinetics of AZD9291 after multiple dosing by assessment of maximum plasma concentration at steady state
Time Frame: PK blood samples are collected multiple times on Cycle 1 Day 8 and Cycle 2 Day 1. Results are based on data cut off of 28 Jan 2016.
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nmol/L
Arm/Group | AZD9291 40mg | AZD9291 80mg
Number analyzed (Participants) | 12 | 12
nmol/L | 303.4 (47.96) | 550.4 (32.35)

9. Primary Outcome: C(ss, Max) of AZ5104 After Multiple Dosing
Description: Pharmacokinetics of AZD9291 metabolites (AZ5104) after multiple dosing by assessment of maximum plasma concentration at steady state
Time Frame: as for outcome 8
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nmol/L
Arm/Group | AZD9291 40mg | AZD9291 80mg
Number analyzed (Participants) | 12 | 13
nmol/L | 29.43 (46.66) | 49.98 (39.73)

10. Primary Outcome: C(ss, Max) of AZ7550 After Multiple Dosing
Description: Pharmacokinetics of AZD9291 metabolites (AZ7550) after multiple dosing by assessment of maximum plasma concentration at steady state
Time Frame: as for outcome 8
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nmol/L
Arm/Group | AZD9291 40mg | AZD9291 80mg
Number analyzed (Participants) | 12 | 13
nmol/L | 25.91 (51.72) | 54.15 (31.34)

11. Primary Outcome: AUC(ss) of AZD9291 After Multiple Dosing
Description: Pharmacokinetics of AZD9291 after multiple dosing by assessment of area under the plasma concentration curve from time zero to the end of the dosing interval
Time Frame: as for outcome 8
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nmol*h/L
Arm/Group | AZD9291 40mg | AZD9291 80mg
Number analyzed (Participants) | 12 | 12
nmol*h/L | 5698 (52.59) | 9570 (35.85)

12. Primary Outcome: AUC(ss) of AZ5104 After Multiple Dosing
Description: Pharmacokinetics of AZD9291 metabolites (AZ5104) after multiple dosing by assessment of area under the plasma concentration curve from time zero to the end of the dosing interval
Time Frame: as for outcome 8
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nmol*h/L
Arm/Group | AZD9291 40mg | AZD9291 80mg
Number analyzed (Participants) | 12 | 13
nmol*h/L | 561.5 (51.74) | 964.7 (37.03)

13. Primary Outcome: AUC(ss) of AZ7550 After Multiple Dosing
Description: Pharmacokinetics of AZD9291 metabolites (AZ7550) after multiple dosing by assessment of area under the plasma concentration curve from time zero to the end of the dosing interval
Time Frame: as for outcome 8
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nmol*h/L
Arm/Group | AZD9291 40mg | AZD9291 80mg
Number analyzed (Participants) | 12 | 12
nmol*h/L | 505.7 (55.23) | 1123 (29.05)

14. Primary Outcome: CL(ss)/F of AZD9291 After Multiple Dosing
Description: Pharmacokinetics of AZD9291 after multiple dosing by assessment of apparent plasma clearance at steady state
Time Frame: as for outcome 8
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: L/h
Arm/Group | AZD9291 40mg | AZD9291 80mg
Number analyzed (Participants) | 12 | 12
L/h | 15.74 (8.532) | 17.67 (6.072)

15. Secondary Outcome: Objective Response Rate (ORR)
Description: Per Response Evaluation Criteria in Solid Tumours (RECIST v1.1) assessed by MRI or CT: Complete Response (CR): Disappearance of all target and non-target lesions and no new lesions; Partial Response (PR): >= 30% decrease in the sum of diameters of Target Lesions (compared to baseline) and no new lesions. ORR is the percentage of patients with at least 1 visit response of CR or PR (according to independent review) that was confirmed at least 4 weeks later, prior to progression or further anti-cancer therapy.
Time Frame: Treatment discontinuation plus 28 days or 12 months after last subject first dose (LSFD). Results are based on data cut off of 2 Nov 2016.
Population: All patients who received at least 1 dose of study treatment and had measurable disease at baseline according to the independent review of baseline imaging data.
Measure: Number (95% Confidence Interval); unit: % of participants
Arm/Group | AZD9291 40mg | AZD9291 80mg
Number analyzed (Participants) | 15 | 16
% of participants | 46.7 [21.27 to 73.41] | 75.0 [47.62 to 92.73]

ADVERSE EVENTS:
Time Frame: AEs from start of study drug until 28 days post treatment discontinuation or 12 months after LSFD. Results are based on data cut off of 2 Nov 2016.
Description: Systematic assessment due to regular investigator assessment at study visits.
Arm/Group | AZD9291 40mg | AZD9291 80mg
Serious Adverse Events (participants affected / at risk) | 3/15 | 5/16
Other Adverse Events (participants affected / at risk) | 15/15 | 16/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AZD9291 40mg (N=15) | AZD9291 80mg (N=16)
Pancreatitis acute (Gastrointestinal disorders) | 0 (0) | 1 (1)
Cholecystitis acute (Hepatobiliary disorders) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Brain oedema (Nervous system disorders) | 0 (0) | 1 (1)
Cerebral artery embolism (Nervous system disorders) | 1 (1) | 0 (0)
Coma (Nervous system disorders) | 0 (0) | 1 (1)
Lethargy (Nervous system disorders) | 1 (1) | 0 (0)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AZD9291 40mg (N=15) | AZD9291 80mg (N=16)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Leukopenia (Blood and lymphatic system disorders) | 4 (10) | 2 (2)
Neutropenia (Blood and lymphatic system disorders) | 2 (6) | 2 (3)
Angina pectoris (Cardiac disorders) | 1 (1) | 0 (0)
Cataract (Eye disorders) | 1 (1) | 0 (0)
Diplopia (Eye disorders) | 1 (1) | 0 (0)
Dry eye (Eye disorders) | 0 (0) | 1 (1)
Eye pruritus (Eye disorders) | 0 (0) | 1 (1)
Eye swelling (Eye disorders) | 1 (1) | 0 (0)
Vision blurred (Eye disorders) | 0 (0) | 1 (1)
Visual acuity reduced (Eye disorders) | 2 (2) | 0 (0)
Xerophthalmia (Eye disorders) | 1 (1) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 2 (2) | 1 (2)
Anal inflammation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 2 (2) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 5 (5) | 11 (19)
Dry mouth (Gastrointestinal disorders) | 3 (3) | 4 (4)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Eructation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 2 (2) | 0 (0)
Gingival pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Haematochezia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 1 (1)
Lip dry (Gastrointestinal disorders) | 0 (0) | 1 (1)
Mouth ulceration (Gastrointestinal disorders) | 1 (3) | 2 (4)
Nausea (Gastrointestinal disorders) | 2 (3) | 2 (2)
Oral mucosal exfoliation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Stomatitis (Gastrointestinal disorders) | 2 (2) | 4 (14)
Toothache (Gastrointestinal disorders) | 1 (1) | 1 (1)
Vomiting (Gastrointestinal disorders) | 6 (9) | 2 (2)
Fatigue (General disorders) | 0 (0) | 2 (2)
Influenza like illness (General disorders) | 1 (1) | 3 (4)
Non-cardiac chest pain (General disorders) | 2 (2) | 3 (5)
Peripheral swelling (General disorders) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 3 (4) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 0 (0) | 1 (1)
Drug-induced liver injury (Hepatobiliary disorders) | 0 (0) | 1 (1)
Jaundice (Hepatobiliary disorders) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 1 (1)
Dermatophytosis (Infections and infestations) | 0 (0) | 1 (2)
Herpes zoster (Infections and infestations) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 1 (1)
Paronychia (Infections and infestations) | 0 (0) | 6 (6)
Pneumonia (Infections and infestations) | 1 (1) | 1 (1)
Respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1) | 2 (2)
Meniscus injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 3 (3) | 1 (1)
Bilirubin conjugated increased (Investigations) | 2 (2) | 0 (0)
Blood bilirubin increased (Investigations) | 1 (1) | 0 (0)
Blood bilirubin unconjugated increased (Investigations) | 1 (1) | 0 (0)
Blood creatinine abnormal (Investigations) | 0 (0) | 1 (1)
Blood creatinine increased (Investigations) | 0 (0) | 2 (2)
Blood sodium decreased (Investigations) | 0 (0) | 1 (1)
Blood urine present (Investigations) | 0 (0) | 1 (1)
Electrocardiogram QT interval abnormal (Investigations) | 0 (0) | 1 (1)
Haemoglobin decreased (Investigations) | 1 (3) | 2 (3)
Neutrophil count decreased (Investigations) | 2 (3) | 5 (10)
Platelet count decreased (Investigations) | 3 (3) | 4 (6)
Red blood cells urine positive (Investigations) | 0 (0) | 2 (2)
White blood cell count decreased (Investigations) | 3 (5) | 6 (16)
Decreased appetite (Metabolism and nutrition disorders) | 3 (3) | 2 (2)
Hypochloraemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 2 (4) | 1 (1)
Hypoproteinaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (3)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2)
Muscle twitching (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Amnesia (Nervous system disorders) | 0 (0) | 1 (1)
Aphasia (Nervous system disorders) | 0 (0) | 1 (1)
Femoral hernia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 2 (3) | 4 (6)
Hyponatraemia (Metabolism and nutrition disorders) | 3 (3) | 1 (1)
Coma (Nervous system disorders) | 0 (0) | 1 (1)
Dysgeusia (Nervous system disorders) | 0 (0) | 1 (1)
Dysstasia (Nervous system disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 3 (3) | 3 (4)
Lethargy (Nervous system disorders) | 1 (1) | 0 (0)
Memory impairment (Nervous system disorders) | 1 (1) | 0 (0)
Nervous system disorder (Nervous system disorders) | 0 (0) | 1 (1)
Neuralgia (Nervous system disorders) | 1 (1) | 0 (0)
Post herpetic neuralgia (Nervous system disorders) | 1 (1) | 0 (0)
Tremor (Nervous system disorders) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 0 (0) | 1 (1)
Soliloquy (Psychiatric disorders) | 1 (1) | 0 (0)
Haematuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Nocturia (Renal and urinary disorders) | 1 (1) | 0 (0)
Proteinuria (Renal and urinary disorders) | 4 (7) | 2 (3)
Urinary retention (Renal and urinary disorders) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (5)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hydrothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Nasal dryness (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2)
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Blister (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 1 (2) | 4 (5)
Dry skin (Skin and subcutaneous tissue disorders) | 5 (5) | 2 (3)
Erythema (Skin and subcutaneous tissue disorders) | 5 (5) | 4 (4)
Nail discolouration (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0)
Onychomadesis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 1 (1) | 3 (4)
Pigmentation disorder (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (3)
Rash (Skin and subcutaneous tissue disorders) | 4 (4) | 1 (2)
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Rash papular (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Rash pruritic (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Skin disorder (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Skin exfoliation (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin fissures (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days